CLINICAL TRIAL: NCT02791204
Title: SPECT/CT Imaging of Skeletal Muscle Perfusion in Healthy Control Subjects and Patients With Peripheral Arterial Disease: Pilot Clinical Study
Brief Title: SPECT/CT Imaging of Skeletal Muscle Perfusion
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Other Study IDs: 1603017342
Record Dates: First submitted 2016-05-25; First posted 2016-06-06 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with PAD: Subjects will undergo resting perfusion imaging of the feet using two separate SPECT/CT systems. Subjects will be injected with a low dose radioisotope. Heated venous blood sampling will be obtained.
  Interventions: Device: SPECT/CT imaging following revascularization procedures
- Controls: Subjects will undergo resting perfusion imaging of the feet using two separate SPECT/CT systems. Subjects will be injected with a low dose radioisotope. In addition to heated venous blood sampling, arterial blood will be continuously sampled from the radial artery for calculation of a blood input function and K1 values for foot angiosomes.
  Interventions: Device: SPECT/CT imaging

INTERVENTIONS:
Device: SPECT/CT imaging following revascularization procedures — Subjects will undergo resting perfusion imaging of the feet using two separate SPECT/CT systems. Subjects will be injected with a low dose radioisotope. Heated venous blood sampling will be obtained.
  Groups: Participants with PAD
Device: SPECT/CT imaging — Subjects will undergo resting perfusion imaging of the feet using two separate SPECT/CT systems. Subjects will be injected with a low dose radioisotope. In addition to heated venous blood sampling, arterial blood will be continuously sampled from the radial artery for calculation of a blood input function and K1 values for foot angiosomes.
  Groups: Controls

SUMMARY:
This study will use SPECT/CT imaging to assess the effect of percutaneous revascularization treatments in patients with Peripheral arterial disease and diabetes mellitus, in whom the disease can progress more quickly than in patients without diabetes.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a progressive atherosclerotic disease of the lower limbs that affects 8 to 10 million Americans, and is more prevalent and progresses more quickly in patients with diabetes mellitus (DM). There is a critical need for a standard non-invasive approach to assess response to treatment by three-dimensional (3D) perfusion to vascular territories of the feet in PAD patients. Assessing the response to treatment is particularly important in DM patients, who suffer from poor distal runoff and often require more distal revascularization to achieve limb salvage.

In this clinical study, the investigators will evaluate lower extremity skeletal muscle perfusion in the feet of healthy controls and PAD patients who are undergoing revascularization using conventional sodium iodide SPECT/CT imaging, as well as dynamic SPECT/CT imaging with a unique cadmium zinc telluride (CZT) system.

Healthy control subjects will be recruited from Yale University and the greater New Haven area. In addition to healthy control subjects, 35 PAD patients with previously diagnosed diabetes will be recruited from Vascular Surgery and Interventional Cardiology at Yale-New Haven Hospital. Patients who are undergoing revascularization procedures will be identified and asked to participate in the imaging study prior to their revascularization procedure and will be imaged once again 1-3 days following revascularization, prior to hospital discharge.

Subjects will undergo resting perfusion imaging of the feet using two separate SPECT/CT systems. They will be injected with a low dose radiotracer. In healthy control subjects, arterial blood will be continuously sampled from the radial artery for calculation of a blood input function and K1 values for foot angiosomes. Additionally, we will sample heated venous "arterialized" blood from a hand vein retrograde to evaluate the potential for heated venous blood in the calculation of a blood input function, thus eliminating the need for arterial access in future PAD patient studies.

ELIGIBILITY:
Inclusion Criteria for Healthy Control Population:

1. At least 18 years of age
2. Normal (0.9-1.2) Ankle Brachial Index

Inclusion Criteria for patients undergoing clinically indicated myocardial perfusion study:

1) At least 18 years of age 2) scheduled for stress myocardial perfusion imaging study for clinically indicated reason

-Inclusion Criteria for PAD Patient Population:

1. At least 18 years of age
2. Evidence of significant obstructive disease for one or multiple lower extremity arteries, as identified by CT angiography, ultrasound, or MR imaging or an abnormal ankle-brachial index or toe-brachial index
3. Previously diagnosed diabetes mellitus (type I or II), based on any of the following criteria: fasting plasma glucose great than 126 mg/dl on 2 separate occasions, glycated hemoglobin (HbA1c) greater than 6.5% on 2 separate occasions, fasting plasma glucose greater than 200 mg/dl 2 hours following an oral glucose tolerance test on 2 separate occasions, or fasting plasma glucose and HbA1c above normal limits on same visit.
4. scheduled for revascularization due to obstructive blood flow in the lower extremities.

Exclusion Criteria for Healthy Control Population:

1. Unable to give informed consent
2. Enrolled in another trial
3. Preexisting medical conditions affecting the vascular system including, but not limited to: Coronary Artery Disease, Peripheral Arterial Disease, diabetes, cancer, hypertension, history of smoking
4. Pregnant or nursing

Exclusion Criteria for PAD Patient Population:

1. Unable to give informed consent or follow-up
2. Enrolled in another trial

Exclusion Criteria for patients undergoing clinically indicated myocardial perfusion study:

1) Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * healthy control subjects will be enrolled for this study.
  * PAD patients with diabetes who are undergoing revascularization procedures
  * patients undergoing clinically indicated myocardial perfusion imaging study
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of effect of percutaneous revascularization treatment measured by change in lower extremity skeletal muscle perfusion before and after treatment using quantitative SPECT/CT imaging of the lower extremities. | patients will be assessed prior to the revascularization procedure (baseline) and a second time 1-3 days following revascularization.
Assessment of lower extremity skeletal muscle perfusion in healthy control subjects compared to patients with peripheral arterial disease and diabetes using quantitative SPECT/CT imaging. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Albert J. Sinusas, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States